CLINICAL TRIAL: NCT04300998
Title: Observational Study of Commercial Chimeric Antigen Receptor T-cell (CAR T) Therapy in Older Patients With Hematologic Malignancies and With an Embedded Pilot Study of Longitudinal Geriatric and Neurocognitive Evaluation
Brief Title: Study of CAR-T Therapy in Older Patients
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-452
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma; Refractory B-Cell Lymphoma; Lymphoma, B-Cell; DLBCL NOS; High-grade B-cell Lymphoma; Multiple Myeloma
Keywords: Lymphoma; CART therapy; relapsed refractory large B-cell lymphoma; High-grade B-cell Lymphoma; DLBCL NOS; Refractory B-Cell Lymphoma; 19-452; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Multiple Myeloma | interventions — Activities of Daily Living; Trail Making Test; Neuropsychological Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- older lymphoma patients: This is a prospective observational cohort where 18 older patients (≥60yo) undergoing CAR T therapy for relapsed refractory high-grade B-cell lymphoma will undergo serial comprehensive geriatric assessment, neurocognitive testing, and quality of life evaluation prior to and following CAR T therapy. The standard follow-up period is one year.
  Interventions: Behavioral: Activities of Daily Living/ADLs; Behavioral: Instrumental Activity of Daily Living; Behavioral: Timed Up and Go; Behavioral: Cognition; Behavioral: Geriatric Depression Scale; Behavioral: Social Support; Behavioral: Brief Test of Attention; Behavioral: Trail Making Test; Behavioral: Controlled Oral Word Association Test; Behavioral: Hopkins Verbal Learning Test-Revised
- older patients with lymphoma and other lymphoid malignancies: This is a prospective observational cohort where 80 older patients (≥60yo) undergoing CAR T therapy for relapsed refractory lymphoma and lymphoid malignancies will undergo comprehensive geriatric assessment, aging biomarker analysis, and quality of life evaluation prior to and following CAR T therapy. The standard follow-up period is one year.
  Interventions: Behavioral: Activities of Daily Living/ADLs; Behavioral: Instrumental Activity of Daily Living; Behavioral: Timed Up and Go; Behavioral: Cognition; Behavioral: Geriatric Depression Scale; Behavioral: Social Support; Behavioral: Brief Test of Attention; Behavioral: Trail Making Test; Behavioral: Controlled Oral Word Association Test; Behavioral: Hopkins Verbal Learning Test-Revised; Other: Blood draw
- older patients with myeloma and other plasma cell disorders: This is a prospective observational cohort where 40 older patients (≥60yo) undergoing CAR T therapy for relapsed refractory plasma cell disorders will undergo
  Interventions: Behavioral: Activities of Daily Living/ADLs; Behavioral: Instrumental Activity of Daily Living; Behavioral: Timed Up and Go; Behavioral: Cognition; Behavioral: Geriatric Depression Scale; Behavioral: Social Support; Behavioral: Brief Test of Attention; Behavioral: Trail Making Test; Behavioral: Controlled Oral Word Association Test; Behavioral: Hopkins Verbal Learning Test-Revised; Other: Blood draw
- older patients with lymphoma: This is prospective observational cohort where 16 older (≥60yo) lymphoma patients with pre-CAR T cognitive impairment.
  Interventions: Behavioral: Activities of Daily Living/ADLs; Behavioral: Instrumental Activity of Daily Living; Behavioral: Timed Up and Go; Behavioral: Cognition; Behavioral: Geriatric Depression Scale; Behavioral: Social Support; Behavioral: Brief Test of Attention; Behavioral: Trail Making Test; Behavioral: Controlled Oral Word Association Test; Behavioral: Hopkins Verbal Learning Test-Revised; Other: Blood draw

INTERVENTIONS:
Behavioral: Activities of Daily Living/ADLs — 7 activities: bathing, dressing, grooming, feeding, walking inside the home, walking outside the home, and bladder and bowel control. Participants get 2 points for each activity that is not limited at all, 1 point for limited a little, and 0 points for limited a lot. Total ADL score ranges from 0 to 14
  Other Names: ADLs
Behavioral: Instrumental Activity of Daily Living — 8 activities: telephone use, doing laundry, shopping, preparing meals, doing housework, handling own medications, handling money and finances, and transportation to visit one's doctor. Participants get 2 points for each activity that can be done without help, 1 point for needing some help, and 0 point for being unable to do. Total iADL score ranges from 0 to16.
  Other Names: iADLS
Behavioral: Timed Up and Go — Participants are asked to get up from the chair, walk 10 feet, turn, and walk back to the char (<10 seconds, 10-20 seconds, >20 seconds)
Behavioral: Cognition — Mini-Cognition test: CDT and 3-word recall
Behavioral: Geriatric Depression Scale — Four yes/no questions regarding patient's psychological status. Score ranges from 0 to 4, and a score of >/=1 is usually indicative of depression.
Behavioral: Social Support — Four 5-point Likert scale questions addressing 4 domains of social support: emotional/ informational, tangible, affectionate, and positive social interaction. Score for each item ranges from 1 to 5, and total score ranges from 4 to 20. A higher score means better social support.
Behavioral: Brief Test of Attention — assess selective auditory attention.
  Other Names: BTA
Behavioral: Trail Making Test — Assesses visual scanning, graphomotor speed, and set shifting.
Behavioral: Controlled Oral Word Association Test — A timed test of verbal fluency
  Other Names: COWAT
Behavioral: Hopkins Verbal Learning Test-Revised — The HVLT-R is a test of verbal learning and recall. Scores obtained are the total number of words: 1) recalled over three trials; 2)recalled after a delay; 3) correctly recognized.
  Other Names: HVLT-R
Other: Blood draw — collection of blood tests
  Groups: older patients with lymphoma; older patients with lymphoma and other lymphoid malignancies; older patients with myeloma and other plasma cell disorders

SUMMARY:
This study is being done to find out how older patients respond to CAR-T cell therapy and how the treatment affects their quality of life. This is a quality of life study and participating in the study does not involve receiving any treatment, other than the standard treatment for participants' disease.

ELIGIBILITY:
Inclusion Criteria:

* are ≥60 years old (all cohorts)
* have pathologically confirmed, relapsed refractory lymphoid malignancy or plasma cell disorder receiving a commercial CAR T-cell product (all cohorts)
* able to speak and understand English (cohort 1 and 4 only)
* have a MoCA score of less than 26 out of 30 during the GA visit by a geriatrician prior to CAR T-cell treatment (cohort 4 only)

Exclusion Criteria:

* Any prior commercial or investigational CAR T therapy (all cohorts)
* Current diagnosis of major Axis I psychiatric disorder (DSM-IV), major depression, bipolar disorder, or schizophrenia, as per medical records or patient report (cohort 1 only)
* History of a neurological disorder, neurodegenerative disease, or traumatic brain injury with loss of consciousness (>60 minutes), as per medical records or patient report (cohort 1 only)
* Current ongoing substance abuse and/or history of substance abuse, as per medical records or patient report (cohort 1 only)
* History of CNS disease (cohort 4 only)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from all oncologists and all transplant physicians at the Memorial Sloan Kettering Cancer Center. Patients are recruited without consideration of gender, country of origin, educational level, or income. There will be no reimbursement or payment toward the participation of this study.
Sampling Method: Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete all required assessment visits prior to disease progression or death | 1 year
  Participants who complete all assessment visits prior to disease progression or death will be considered as a success for a feasibility endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lin, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org